CLINICAL TRIAL: NCT07063381
Title: Effect of Low-frequency Electrical Stimulation of the Auricular Branch of the Vagus Nerve on Cognitive Function in Patients With Atrial Fibrillation
Brief Title: Low-frequency Electrical Stimulation for Cognitive Enhancement in Atrial Fibrillation
Acronym: LESCAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bakulev Scientific Center of Cardiovascular Surgery (Other Government)
Collaborators: Lobachevsky University (Unknown)
Responsible Party: Principal Investigator, Vladimir A Shvartz, MD, Principal Investigator, Bakulev Scientific Center of Cardiovascular Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0034.2025; H-465-99_2025-2027 (Other: Lobachevsky State University of Nizhny Novgorod)
Record Dates: First submitted 2025-06-23; First posted 2025-07-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Function Abnormal; Atrial Fibrillation (AF)
Keywords: transcutaneous vagus nerve stimulation; vagus nerve stimulation; atrial fibrillation; auricular vagus nerve stimulation; cognitive functions; memory; executive functions; information processing speed; modulation of parasympathetic activity; neuroplasticity; neurotrophic factors; cerebral blood flow; inflammatory cytokines
MeSH Terms: conditions — Cognition Disorders; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A randomized double-blind controlled trial in two groups (1:1)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Active Comparator): Active stimulation will be carried out using the tVNS device with an ear clip attached to the tragus of the left ear at a frequency of 20 Hz, 250 μs at a current slightly below the discomfort threshold. The device's operating mode is active therapeutic.
  Interventions: Device: tVNS
- Sham tVNS (Sham Comparator): Fictitious stimulation will be carried out using the tVNS device with an ear clip attached to the tragus of the left ear at a frequency of 20 Hz, 250 μs at a current slightly below the discomfort threshold. The device's operating mode is research mode.
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tVNS — tVNS will be performed daily after workouts for 60 minutes over a period of 6 months.

SUMMARY:
Cognitive function in patients with atrial fibrillation (AF) is often impaired due to the complex influence of various factors (cerebral hypoperfusion, neurodegeneration, microemboli, hypertension, chronic inflammation). This leads to impairment of cognitive functions, including attention, memory, executive functions, and speed of information processing. The search for affordable and safe methods to maintain or improve cognitive function in this group of people is an urgent task of modern medicine. One of the promising approaches is percutaneous low-frequency electrical stimulation of the auricular branch of the vagus nerve (transcutaneous Vagus Nerve Stimulation - tVNS).

The auricular (auricular) branch of the vagus nerve is a peripheral branch of the vagus nerve innervating the skin of the auricle in the area of the tragus and the inner part of the external auditory canal. The tVNS engages the sensory fibres of the vagus nerve and thus mimics the sensory input to the brainstem, forming the so-called auriculo-vagal afferent pathway. Since these fibres project directly to the nucleus of the solitary pathway (solitary tract), which, in turn, has direct and indirect projections to the nuclei providing noradrenergic, endorphinergic and serotoninergic fibres in various parts of the brain regulating systemic indices of cardiovascular, respiratory and immunological functions, the organism's response to stimulation of the auricular branch of the vagus nerve is systemic in nature.

Stimulation of this nerve can modulate central nervous system (CNS) activity, affecting processes related to memory, attention and emotional state. Mechanisms of action of tVNS include modulation of parasympathetic activity, enhancement of neuroplasticity through increased expression of neurotrophic factors (e.g., BDNF), improvement of cerebral blood circulation, and regulation of neuroinflammation (reduction of proinflammatory cytokines).

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years,
* Permanent form of AF,
* Severe and mild cognitive impairment (<26 points on the MoCA-8 test),
* The possibility of regular repeat visits for 6 months.

Exclusion Criteria:

* Atrioventricular blockade of 2-3 degree,
* Expressed sinus bradycardia with resting heart rate < 40 bpm
* Any oncological diseases,
* Severe chronic liver and kidney pathology,
* Chronic viral infections.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamics of neural activity of the brain. | This parameter will be assessed at the beginning of the study (initially) and at the end of the study (6 months) in the active and fictitious stimulation groups.
  Changes in the characteristics of time-frequency analysis of the neural activity of the brain associated with the performance of a cognitive task.

SECONDARY OUTCOMES:
Reaction Time (RT) Changes & EEG Correlates | This parameter will be assessed at the beginning of the study (initially) and at the end of the study (6 months) in the active and fictitious stimulation groups.
  Changes in reaction time (RT) during the perception and classification of ambiguous visual stimuli (Necker cubes) by a patient. The test is conducted with simultaneous EEG recording during the visual task (determining the orientation of the Necker cube - right-oriented or left-oriented configuration).
  The presentation of ambiguous stimuli, such as the Necker cube, leads to an increase in reaction time due to the need to resolve perceptual conflict and make decisions under uncertainty. Parallel EEG recording reveals specific neural correlates of this process (N200 - conflict, P300 - decision/classification, frontal theta - cognitive control, gamma - perceptual reorganization), which are directly related to the observed changes in reaction speed. Analysis of these EEG markers together with RT provides deep insight into brain dynamics during the processing of ambiguous information.
Attention Level Changes & Error Rates | This parameter will be assessed at the beginning of the study (initially) and at the end of the study (6 months) in the active and fictitious stimulation groups.
  Changes in the level of attention during the perception and classification of ambiguous visual stimuli (Necker cubes) by a patient. The test is conducted with simultaneous EEG recording during the visual task (determining the orientation of the Necker cube - right-oriented or left-oriented configuration). The frequency of actual errors (incorrect reporting) is assessed.
  The presentation of ambiguous stimuli, such as the Necker cube, requires an increased level of attention (especially executive control), reflected in specific EEG patterns (theta, N2, P3). The primary sources of errors are perceptual instability (switches during response) and unresolved conflict/uncertainty. Analysis of EEG (ERN/Pe) allows studying the process of error detection and correction itself.
Dynamics of the cognitive test MoCA-8 (Montreal Cognitive Assessment). | This parameter will be assessed at the beginning of the study (initially) and at the end of the study (6 months) in the active and fictitious stimulation groups.
  Changes in the MoCA-8 score. Scores on the MoCA-8 test range from 0 to 30, where a score <26 may indicate cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Bakulev National Medical Research Center for Cardiovascular Surgery, Moscow
  - Neurodynamics and Cognitive Technologies Research Laboratory of the Neuroscience Research Institute, Nizhny Novgorod

IPD SHARING:
Plan to Share IPD: No